CLINICAL TRIAL: NCT03107741
Title: Effectiveness of Tai Chi Training to Alleviate Metabolic Syndrome in Abdominal Obese Older Adults: A Randomized Controlled Trial
Brief Title: Effectiveness of Tai Chi Training on Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Angus Yu (Other)
Responsible Party: Sponsor-Investigator, Angus Yu, Research Assistant, The Hong Kong Polytechnic University
Organization: The Hong Kong Polytechnic University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Tai Chi and Metabolic Syndrome
Record Dates: First submitted 2017-04-05; First posted 2017-04-11 (Actual); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: Metabolic Syndrome
Keywords: Metabolic Syndrome; Waist circumference; Blood pressure; Triglyceride; HDL cholesterol
MeSH Terms: conditions — Metabolic Syndrome | interventions — Tai Ji

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (3):
- Passive Control (No Intervention): Subjects in this group will not receive any intervention.
- Conventional Exercise (Placebo Comparator): Subjects in this group will receive three 1-hour conventional exercise training sections per week for 12 weeks
  Interventions: Other: Conventional Exercise
- Tai Chi (Active Comparator): Subjects in this group will receive three 1-hour tai chi training sections per week for 12 weeks
  Interventions: Other: Tai Chi

INTERVENTIONS:
Other: Conventional Exercise — Subjects in this group will receive three 1-hour conventional exercise training sections per week for 12 weeks
  Arms: Conventional Exercise
Other: Tai Chi — Subjects in this group will receive three 1-hour tai chi training sections per week for 12 weeks
  Arms: Tai Chi

SUMMARY:
Metabolic syndrome (MetS) is a serious public health problem in Hong Kong and worldwide. Older adults, the age group with the highest prevalence of MetS, may prefer specific exercise modalities that are suitable for their regular participation to manage MetS. This project aims to evaluate the effectiveness of Tai Chi, a very suitable exercise for older adults, to alleviate MetS in older population

DETAILED DESCRIPTION:
PURPOSE/OBJECTIVE: Metabolic syndrome (MetS) is a serious public health problem in Hong Kong and worldwide. Older adults, the age by specific exercise modalities that are suitable for regular participation. This project aims to evaluate the effectiveness of Tai Chi to alleviate MetS in older population.

DESIGN & METHODS: This study is a three-arm assesscer blinded randomized controlled trial. Older adults aged 50 years or above with abdominal obesity will be randomly assigned to passive control, active control and Tai Chi groups. Subjects assigned to Tai Chi and active control groups will receive a 12-week intervention of Tai Chi and generic fitness, respectively. No intervention will be given to the passive control group. Outcome measures including waist circumference, blood pressure, blood glucose, triglyceride and high density lipoprotein-cholesterol will be assessed at baseline, post-intervention and follow-up (6 months after the end of intervention) assessments in all groups.

HYPOTHESES: We hypothesize that: 1) improvements of waist circumference and other indicators of MetS are found in Tai Chi group but not in passive control group and 2) improvements of waist circumference and other indicators of MetS are more profound in Tai Chi group than active control group.

ELIGIBILITY:
Inclusion Criteria:

* Ethnic Chinese
* Abdominal Obese: Meeting the defined criteria of International Diabetes Federation (IDF) and National Cholesterol Education Program (NCEP) for abdominal obesity using Asian-specific cut off (waist circumference ≥ 90 cm for male; ≥ 80 cm for female)

Exclusion Criteria:

* Regularly practice moderate-intensity exercise or tai chi (>3 times a week of >30-min/ session)
* Serious medical and somatic condition that prevent participation in generic fitness/Tai Chi exercise
* Serious chronic diseases known to affect mobility (eg. Neurological diseases, musculoskeletal disorder and autoimmune diseases)
* Under treatment for serious chronic diseases (eg. Cancer treatment)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 543 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Waist circumference | Immediately after completion of the 12-week intervention
  Waist circumference will be measured midway between the lowest rib and the superior border of the iliac crest using an inelastic measuring tape on the bare skin to the nearest 0.1 cm. Measurement will be performed at the end of normal expiration.
Waist circumference | 6 months after the completion of intervention
  Waist circumference will be measured midway between the lowest rib and the superior border of the iliac crest using an inelastic measuring tape on the bare skin to the nearest 0.1 cm. Measurement will be performed at the end of normal expiration.

SECONDARY OUTCOMES:
Remission of central obesity | Immediately after completion of the 12-week intervention and 6 months after the completion of intervention
  The percentage of subjects that no longer diagnosed with central obesity according to the criterion of International Diabetes Federation (IDF) and National Cholesterol Education Program (NCEP) for abdominal obesity using Asian-specific cut off (waist circumference ≥ 90 cm for male; ≥ 80 cm for female).
Blood triglyceride | Immediately after completion of the 12-week intervention and 6 months after the completion of intervention
  Biochemical measurements will be performed in venous blood samples collected after overnight fast. Subjects will come to our laboratory after an overnight (≥ 8 hours) fasting. Subjects will sit in a quiet environment for 15 minutes prior to blood collection. Venous blood will be drawn from an antecubital vein in the forearm by a licensed phlebotomist. The level of blood triglyceride will be measured by an accredited medical laboratory.
High density lipoprotein-cholesterol | Immediately after completion of the 12-week intervention and 6 months after the completion of intervention
  Biochemical measurements will be performed in venous blood samples collected after overnight fast. Subjects will come to our laboratory after an overnight (≥ 8 hours) fasting. Subjects will sit in a quiet environment for 15 minutes prior to blood collection. Venous blood will be drawn from an antecubital vein in the forearm by a licensed phlebotomist. The level of HDL-cholesterol will be measured by an accredited medical laboratory.
Fasting blood glucose | Immediately after completion of the 12-week intervention and 6 months after the completion of intervention
  Biochemical measurements will be performed in venous blood samples collected after overnight fast. Subjects will come to our laboratory after an overnight (≥ 8 hours) fasting. Subjects will sit in a quiet environment for 15 minutes prior to blood collection. Venous blood will be drawn from an antecubital vein in the forearm by a licensed phlebotomist. The level of blood glucose will be measured by an accredited medical laboratory.
Systolic blood pressure | Immediately after completion of the 12-week intervention and 6 months after the completion of intervention
  Blood pressure measurement will be measured on the right arm after a 5-minute seated rest using the Datascope Accutorr Plus BP Monitor. Systolic and diastolic blood pressure will be obtained over brachial artery region with the arm supported at heart level using appropriate sized cuff. The average of two measurements taken within one minute interval will be recorded for analysis.
Diastolic blood pressure | Immediately after completion of the 12-week intervention and 6 months after the completion of intervention
  Blood pressure measurement will be measured on the right arm after a 5-minute seated rest using the Datascope Accutorr Plus BP Monitor. Systolic and diastolic blood pressure will be obtained over brachial artery region with the arm supported at heart level using appropriate sized cuff. The average of two measurements taken within one minute interval will be recorded for analysis.
Bodyweight | Immediately after completion of the 12-week intervention and 6 months after the completion of intervention
  A calibrated electronic digital weighing scale with a capacity from 0.05kg to 150kg (± 0.05kg accuracy) will be used to weigh the subjects.
Body mass index | Immediately after completion of the 12-week intervention and 6 months after the completion of intervention
  A calibrated electronic digital weighing scale with a capacity from 0.05kg to 150kg (± 0.05kg accuracy) will be used to weigh the subjects. A stadiometer (Holtain Ltd., UK) with 200 cm limit and ± 0.01 cm accuracy will be used to measure body height. The BMI will be calculated from the body weight and height.

CONTACTS AND LOCATIONS:
Overall Officials: Parco MF Siu, PhD, Principal Investigator — The University of Hong Kong
Locations (2):
- Hong Kong (2):
  - The Hong Kong Polytechnic University, Hong Kong
  - The University of Hong Kong, Hong Kong

REFERENCES:
- [Derived] Siu PM, Yu AP, Chin EC, Yu DS, Hui SS, Woo J, Fong DY, Wei GX, Irwin MR. Effects of Tai Chi or Conventional Exercise on Central Obesity in Middle-Aged and Older Adults : A Three-Group Randomized Controlled Trial. Ann Intern Med. 2021 Aug;174(8):1050-1057. doi: 10.7326/M20-7014. Epub 2021 Jun 1. PMID 34058100